CLINICAL TRIAL: NCT06679725
Title: Effects of Wild Ginseng Extract on Exercise Performance, Cognitive Function, and Fatigue Recovery Using College Students: a Randomized Cross-Over, Placebo-Controlled, and Double-Blind Study
Brief Title: The Investigators Conducted a Study to Examine the Impact of Wild Ginseng Extract (WG) on Exercise Performance, Cognitive Function, and Fatigue Recovery Among Twelve Healthy Adult Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University San Antonio (Other)
Responsible Party: Principal Investigator, Dr. Suk H. Lee, Professor of Health and KInesiology, Texas A&M University San Antonio
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Wild Ginseng Extract; 11072014 (Other: Korea Food Research Institute)
Record Dates: First submitted 2024-10-26; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Ginseng; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Asian ginseng

STUDY DESIGN:
Intervention Model Description: This study is a double-blind, placebo-controlled crossover experiment with two trials (WG and placebo) separated with 2-week wash-out period.
Who Masked: Participant, Investigator
Masking Description: Double blind study using identical-looking package. The taste of the beverage was very similar for both WG and placebo (based on food survey)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wild ginseng extract (Experimental): The ginseng used in this study is a commercially manufactured standardized 140 ml liquid package and approved for safety. The drink contains 0.25% of wild ginseng extract and other ingredients while the placebo is manufactured to be identical in appearance (brown color, calorie (30.23 Kcal), taste, and content). The placebo utilized in the study consisted of the same ingredients as the treatment drink, with the exception of 0.25% wild ginseng extract.
  Interventions: Dietary Supplement: Wild ginseng extract
- Placebo (Placebo Comparator): The placebo utilized in the study consisted of the same ingredients as the treatment drink, with the exception of 0.25% Korean wild Ginseng Extract. This was achieved by incor-porating 0.25% scented ginseng and 0.06% caramel coloring (Table 1).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wild ginseng extract — This ginseng extract was manufactured and provided by the Korea Food Research Institute (sponsor). It is extracted from red ginseng. Red ginseng is generally considered to have greater biological effects and fewer side effects than white or fresh ginseng.
  Other Names: Ginseng extract
  Arms: Wild ginseng extract
Dietary Supplement: Placebo — The placebo utilized in the study consisted of the same ingredients as the treatment drink, with the exception of 0.25% Korean wild Ginseng Extract. This was achieved by incor-porating 0.25% scented ginseng and 0.06% caramel coloring
  Arms: Placebo

SUMMARY:
The goal of this clinical trial was to learn if Wild Ginseng extract (WG) influences exercise performance, cognitive function, and fatigue recovery from the exercise.

The main questions to answer were:

* Does WG improve exercise performance?
* Does WG improve cognitive function?
* Does WG facilitate recovery from the exercise?

The investigators will compare WG to a Placebo (a look-alike substance that contains no substance) to see if WG works.

Participants will:

* Take WG or a Placebo every day for 7 days with a 2-week wash-out (It is a specific time frame. During this time, certain substances are removed from the body).
* Visit the laboratory a total of five times for the tests, including one pre-familiarization (to be familiar with the exercise and other procedures)

DETAILED DESCRIPTION:
Dietary supplements are used by athletes worldwide. In the United States, the Dietary Supplement Health Education Act has defined dietary supplements as something added to the diet, mainly vitamins, minerals, protein, herbs or botanicals, and metabolites/constituents/extracts, or a combination of any of these ingredients. In the realm of sports performance enhancement, the quest for safe and effective ergogenic aids continues to evolve. With the evolving landscape of supplementation, a significant portion of the Americans tends to favor very specific supplements.

Among the plethora of natural substances garnering attention, wild ginseng extract emerges as a compelling candidate. Ginseng is widely used for its promising healing and restorative properties as well as for its possible tonic effect in traditional medicine and has recently become a popular supplement in Western Countries. There are a multitude of variations among ginseng: among those, Korean ginseng is most notable for its efficacy. To date there have been numerous studies utilizing Korean ginseng attempting to establish an increase in either sports performance, cognitive function, or fatigue recovery. The use of ginseng thus far has not proved much success in the realm of performance enhancement. Conversely, notable achievements have been observed in the realms of cognitive enhancement and fatigue mitigation. The wild ginseng extract has exhibited promising results in ameliorating psychomotor performance and mitigating the effects of chronic fatigue associated with various pathological conditions.

Some issues arise from previous studies of ginseng use as an ergonomic aid. First are the inadequate sample sizes that are being utilized. Secondly are the varying dosages that are being used throughout the study. The issues that arise with all previous studies are the varying doses along with inadequate sample sizes. The limitations of previous investigations lie predominantly in their emphasis on chronic effects, or their exclusive focus on specific domains such as endurance sports and cognitive function. Consequently, there remains a notable scarcity of research delving into the acute impacts of wild ginseng extract on exercise performance, cognitive function, and fatigue recovery. Therefore, the primary objective of this study was to elucidate the effects of wild ginseng extract on exercise performance, cognitive function, and fatigue recovery.

This study is a double-blind, placebo-controlled crossover experiment with two trials (WG and placebo). Twelve healthy adult males (age=31±6.86 years) were randomly assigned to either WG or placebo groups with 2-week wash-out period. After a brief explanation of procedures, exercises, risks, and benefits associated with the study, each participant gave written consent before participation. The study was approved by the College's Institutional Review Board. Participants completed a questionnaire before the initiation of the experiment. Any of the participants who had any health issues, injuries, metabolic, cardiovascular, pulmonary disease, or intake of medication and or herbal supplementation were excluded from the trials.

Before the test, The investigators had a pre-familiarization that was conducted 3-5 days prior to the experiment. During the pre-familiarization, The investigators conducted a VO2 max test, body composition measurements, and cognitive function test. Body Composition. Body weight, height, percentage of body fat, blood pressure (mmHg), and heart rate (beats/min) were assessed. Body weight and height (weight in kilograms, height in meters) were measured using a wall stadiometer (PAT #290237, Novel Products, USA). Body fat (kg) was measured by skin fold (PAT#3,008,239, Beta Technology, USA). Blood pressure (mmHg) was measured using a blood pressure gauge (BP791IT, Omron, Japan). Heart rate (beats/min) was assessed by using a heart rate monitor (S120, Polar, USA). After the pre-familiarization, the experiments began. A Korean wild ginseng extract drink or placebo was given 90 minutes before the cycling exercise began. Power, strength, and cognitive function tests were conducted before, during, and after the experiment.

Composition of WG and Placebo Ingredient Ginseng Drink (%) Placebo (%) Korea Wild Ginseng Extract 0.25 0.00 Soy Powder 1.5 1.5 Almond Paste 1.5 1.5 Isomaltooligosaccharide 1.0 1.0 Fructooligosaccharide 0.75 0.75 Refined Salt 0.95 0.95 Scented Almond 0.05 0.05 Xanthan Gum 0.95 0.95 Sodium Bicarbonate 0.95 0.95 Soybean Extract 0.5 0.5 Water 93.15 93.15 Scented Ginseng 0.00 0.25 Caramel Coloring 0.00 0.06

VO2 max test: The participants were initially tested on a cycle ergometer to determine their maximal aerobic capacity (VO2 max) to accurately prescribe exercise intensities for endurance performance. During the VO2 max test, the participants exercised on cycle ergometer (894E, Monark, Sweden) with an initial work rate equal to 60 W and a pedaling rate of 60 revolutions per minute (rpm) for 2 minutes. Thereafter, the work rate increased by 30W every 2 minutes until the participant reached exhaustion, which was determined when participants met at least 2 of the following conditions: (a) inability to keep up the pedaling rate of 60 rpm for more than 5 seconds with verbal encouragement, (b) respiratory exchange ratio (RER) 1.10, (c) rating of perceived exertion (RPE) ≧19 (Borg 6-20 scale), or (d) volitional fatigue.

Cycling exercise: The participants performed the cycling exercise to assess endurance performance for 30 minutes at 70-75% of VO2 max. The cycle ergometer (984E, Monark, Sweden) was used to perform the cycling exercise.

Exercise Performance measurements Power: Power (Watts/kg) was evaluated by peak (average) power test using automatic Powercycle (Powercycle, USA). The participants performed a 2-minute warm-up by cycling at 100 to 120 repetitions per mins (rpm) with a power of 100 to 120 Watts. They performed four bouts of maximal acceleration for approximately 3 to 4 seconds on a verbal command with standardized encouragement. Data was recorded for 6.5 crank revolutions. The length of seat height was selected by each participant.

Strength: Isometric knee extensor and flexor strength (kg) was measured by a muscle testing system (Lafayette, USA). The participants sat on the table in supine position, and the knee and hip are positioned 90 degrees. The participants were instructed to remain seated and place both hands on the table. The dynamometer force pad was placed proximal to the ankle joint, and the knee extensor strength was quantified in pound force. All participants performed two maximal trials for 3 to 5 seconds with a 30 second rest interval. The higher value of two trials was recorded with normalized as a direct percentage of body weight (%BW).

Endurance performance: The participant performed the 10-mile time trial to assess endurance performance (second) using cycle ergometer. The cycle ergometer (984E, Monark, Sweden) was used to perform the time trial cycling. The workload was standardized for each participant by setting the resistance to achieve 70% VO2 max. Participants received standard encouragement to complete the time trial as quickly as possible and the time to complete the 10-mile distance was recorded.

Blood Analysis Glucose, IL-6, myoglobin, and total antioxidant capacity (TAC) were measured using about 2.5- 3 ml of blood withdrawn from an antecubital vein before, during, and after the cycling performances. The total volume of blood withdrawn per test was less than 34 ml. Therefore, total amount of blood withdrawn for all tests was less than 136 ml over the 44 days of experimental period (34 ml x 4 tests = 136 ml) A trained phlebotomist used the same standardized procedure used in doctors' offices and labs to collect blood. All blood samples were drawn into a tube containing ethylenediamine tetra-acetic acid (EDTA) to prevent coagulation. The blood was centrifuged, and the upper layer of plasma was transferred into a conical tube and stored at -20°C. Plasma lactate was then analyzed by lactic dehydrogenase enzymatic method (Sigma, USA). Serum was analyzed for glucose, IL-6, myoglobin, and total antioxidant capacity (TAC). Glucose level was analyzed by oxidase/Trinder endpoint method (Fisher, USA). IL-6 was analyzed by commercially available enzyme-linked immunosorbent assay (ELISA, EMD Millipore, Germany). Myoglobin was analyzed by enzyme immunoassay (ELISA, Biocheck, USA). Total antioxidant capacity (TAC) was analyzed using an antioxidant assay kit. All measurements were performed in duplicate.

Cognitive Performance To assess cognitive function, psychomotor vigilance task (PVT) and delayed-match-to-sample task (DMS) were taken before and after each exercise. The PVT test is composed of 40 trials for 5 minutes to assess mean reaction time (msec). The DMS was taken 20 minutes with 20 trials to assess memory.

Fatigue Fatigue rates were measured utilizing a rate of perceived exertion (RPE), scale of muscle soreness, and a fatigue questionnaire that was provided.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects (age from 18-30 years old) that have no health problems, injuries, metabolic, cardiovascular, or pulmonary disease.
* No history of taking prescription medications or herbals

Exclusion Criteria:

• Having health problems, injuries, metabolic, cardiovascular, or pulmonary disease.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Peak and average power outputs (Watts/kg) | through study completion, an average of 3 months
  The participants performed a 2-minute warm-up by cycling at 100 to 120 revolutions per minute with a power of 100 to 120 Watts using an automatic Powercycle (Powercycle, USA). They performed four bouts of maximal acceleration for approximately 3 to 4 seconds on a verbal command with standardized encouragement. Data was recorded for 6.5 crank revolutions. The length of seat height was selected by each subject.
Strength (kg) | through study completion, an average of 3 months
  Isometric knee extensor and flexor strength were measured by a muscle testing system (Lafayette, USA). The participants sat on the table in supine position, and the knee and hip are positioned 90 degrees. The participants were instructed to remain seated and place both hands on the table. The dynamometer force pad was placed proximal to the ankle joint, and the knee extensor strength was quantified in pound force. All participants performed two maximal trials for 3 to 5 seconds with a 30-second rest interval. The higher value of the two trials was recorded.
Endurance (time: minutes and seconds) | through study completion, an average of 3 months
  The participants performed the 10-mile time trial to assess endurance performance (second) using a cycle ergometer. The cycle ergometer (984E, Monark, Sweden) was used to perform the time trial cycling. The workload was standardized for each subject by setting the resistance to achieve 70% VO2 max (maximal oxygen consumption measured during 1st lab visit). Subjects received standard encouragement to complete the time trial as quickly as possible and the time (minute and second) to complete the 10-mile distance was recorded.
Cognitive function (psychomotor vigilance task (PVT): msec) | through study completion, an average of 3 months
  The PVT test is composed of 40 trials for 5 minutes to assess mean reaction time (msec). Participants were instructed to attend to a small, fix point at the center of a computer screen for 2 s (sec) and then respond via button press as rapidly as possible between 100 milliseconds (msec) and 500 msec upon detection of a msec counter on the screen. The stimulus was presented at random time intervals between 2 and 10 s. The final counter values corresponded to the participant's reaction time. Response success (within a range of 100-500 msec) or failure (< 100 msec or> 500 msec) was displayed on the window screen for
  1 s, thus providing feedback for reaction time (msec) and data were stored on the computer as average reaction time (msec) and the number of correct trials. PVT took approximately 5 min and consisted of 45 trials.
Cognitive function (match-to-sample memory task (DMS): msec and number of correct trials) | through study completion, an average of 3 months
  With an initial key press, participants viewed and studied a 5× 5 grid of brightly colored yellow and red squares with a unique pattern on a computer screen. After another key press, the stimulus disappeared, and the screen became blank through a 6 s-delay period, and then two stimuli were presented on the screen (a "match" and "non-match"). Participants were asked to indicate which stimulus was the correct "match" with a key press and to respond as quickly and as accurately as possible, thus providing feedback for either "correct" or "incorrect" trial in 1 s. After completing 30 trials for 5-6 min, the final counter values were stored on the computer as average study time (msec), memory retrieval latency (msec), and the number of correct trials.
Fatigue recovery (scale (6-20) and fatigue questionnaire) | through study completion, an average of 3 months
  Fatigue recovery rates were measured utilizing a rate of perceived exertion (RPE), a scale of muscle soreness, and a fatigue questionnaire that was provided.
  The Borg RPE scale rates exertion from a scale of 6 (no exertion) to 20 (maximum effort). A rating between 12 to 14 typically reflects a moderate or somewhat hard level of intensity.

SECONDARY OUTCOMES:
Maximal aerobic capacity (VO2 max) (ml/kg/min) | One day: one time at the beginning of the study (1st visit).
  To accurately prescribe exercise intensities for endurance performance. During the VO2 max test, the subjects exercised on a cycle ergometer (894E, Monark, Sweden) with an initial work rate equal to 60 W and a pedaling rate of 60 revolutions per minute (rpm) for 2 minutes. After that, the work rate increased by 30 Watts every 2 minutes until the subject reached exhaustion, which was determined when subjects met at least 2 of the following conditions: (a) inability to keep up the pedaling rate of 60 rpm for more than 5 seconds with verbal encouragement, (b) respiratory exchange ratio (RER) 1.10, (c) rating of perceived exertion (RPE) ≧19 (Borg 6-20 scale), or (d) volitional fatigue.
Height (cm) | One day: one time at the beginning of the study (1st visit).
  The height was measured using a wall stadiometer (PAT #290237, Novel Products, USA).
Body weight (kg and lb) | One day: one time at the beginning of the study (1st visit).
  Body weight was measured using a standard scale.
Heart rate (beats per mins (BPM)) | One day: one time at the beginning of the study (1st visit).
  Heart rate was assessed by using a heart rate monitor (S120, Polar, USA)
Body fat (%) | One day: one time at the beginning of the study (1st visit).
  Body fat was measured by skin fold (PAT#3,008,239, Beta Technology, USA). Estimate body fat % based on measurements of subcutaneous fat. Measurements are taken on the right side of body. Caliber needs to be perpendicular to the site analyzed. The participant must relax the muscle group that is being assessed. When skin fold is pinched, the practitioner should be taking reading at the middle of the pinched skin, not apex or base. Wait 1 to 2 seconds after releasing caliber, record closest 0.5mm. Retake each site in order to obtain accurate readings.
  Male measurements: Chest, abdominal, and thigh. Female measurements: Tricep: suprailiac, and thigh. Body Fat Percentage = (27 x sum of skinfold sites) divided by bodyweight (lb.)
Blood pressure (mmHg) | One day: one time at the beginning of the study (1st visit).
  Blood pressures (systolic and diastolic) were measured using a blood pressure gauge (BP791IT, Omron, Japan).
Blood Analysis (Glucose (mg/dL)) | Two days (two separate visits). Total 7 time points (0, 100, 140, right after time trial, 30, 60, and 120 mins after time trial test) mins) during the each trail. 7 time points x 2 trials = 14 times.
  The blood glucose was measured using about 2.5- 3 ml of blood withdrawn from an antecubital vein before, during, and after the cycling performances. Glucose level was analyzed by oxidase/Trinder endpoint method (Fisher, USA). The total volume of blood withdrawn per test was less than 34 ml. All blood samples were drawn into a tube containing ethylenediamine tetra-acetic acid (EDTA) to prevent coagulation. The blood was centrifuged, and the upper layer of plasma was transferred into a conical tube and stored at -20°C.
Blood Analysis (Interleukin-6 (IL-6: pg/mL)) | Two days (two separate visits). Total 7 time points (0, 100, 140, right after time trial, 30, 60, and 120 mins after time trial test) mins) during the each trail. 7 time points x 2 trials = 14 times.
  IL-6 was analyzed by commercially available enzyme-linked immunosorbent assay (ELISA, EMD Millipore, Germany). It was measured using about 2.5- 3 ml of blood withdrawn from an antecubital vein before, during, and after the cycling performances. The total volume of blood withdrawn per test was less than 34 ml. All blood samples were drawn into a tube containing ethylenediamine tetra-acetic acid (EDTA) to prevent coagulation. The blood was centrifuged, and the upper layer of plasma was transferred into a conical tube and stored at -20°C.
Blood Analysis (Myoglobin (mcg/L)) | Two days (two separate visits). Total 7 time points (0, 100, 140, right after time trial, 30, 60, and 120 mins after time trial test) mins) during the each trail. 7 time points x 2 trials = 14 times.
  Myoglobin was analyzed by enzyme immunoassay (ELISA, Biocheck, USA). It was measured using about 2.5- 3 ml of blood withdrawn from an antecubital vein before, during, and after the cycling performances. The total volume of blood withdrawn per test was less than 34 ml. All blood samples were drawn into a tube containing ethylenediamine tetra-acetic acid (EDTA) to prevent coagulation. The blood was centrifuged, and the upper layer of plasma was transferred into a conical tube and stored at -20°C
Blood Analysis (Total antioxidant capacity (TAC): nM) | Two days (two separate visits). Total 7 time points (0, 100, 140, right after time trial, 30, 60, and 120 mins after time trial test) mins) during the each trail. 7 time points x 2 trials = 14 times.
  Total antioxidant capacity (TAC) was analyzed using an antioxidant assay kit. All measurements were performed in duplicate. It was measured using about 2.5- 3 ml of blood withdrawn from an antecubital vein before, during, and after the cycling performances. Glucose level was analyzed by oxidase/Trinder endpoint method (Fisher, USA). The total volume of blood withdrawn per test was less than 34 ml. All blood samples were drawn into a tube containing ethylenediamine tetra-acetic acid (EDTA) to prevent coagulation. The blood was centrifuged, and the upper layer of plasma was transferred into a conical tube and stored at -20°C.
Blood Analysis (Cortisol (ng/ml)) | Two days (two separate visits). Total 7 time points (0, 100, 140, right after time trial, 30, 60, and 120 mins after time trial test) mins) during the each trail. 7 time points x 2 trials = 14 times.
  The cortisol was analyzed by commercially available enzyme-linked immunosorbent assay (ELISA, DRG, USA). It was measured using about 2.5- 3 ml of blood withdrawn from an antecubital vein before, during, and after the cycling performances. The total volume of blood withdrawn per test was less than 34 ml. All blood samples were drawn into a tube containing ethylenediamine tetra-acetic acid (EDTA) to prevent coagulation. The blood was centrifuged, and the upper layer of plasma was transferred into a conical tube and stored at -20°C.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University-San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The enrollment of this study was completed in 2016.

REFERENCES:
- [Background] Zhu J, Xu X, Zhang X, Zhuo Y, Chen S, Zhong C, Liu M, Wang Z. Efficacy of ginseng supplements on disease-related fatigue: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Jul 1;101(26):e29767. doi: 10.1097/MD.0000000000029767. PMID 35776997
- [Background] Bentler SE, Hartz AJ, Kuhn EM. Prospective observational study of treatments for unexplained chronic fatigue. J Clin Psychiatry. 2005 May;66(5):625-32. doi: 10.4088/jcp.v66n0513. PMID 15889950
- [Background] Kennedy DO, Scholey AB, Wesnes KA. Dose dependent changes in cognitive performance and mood following acute administration of Ginseng to healthy young volunteers. Nutr Neurosci. 2001;4(4):295-310. doi: 10.1080/1028415x.2001.11747370. PMID 11842896
- [Background] Scholey AB, Kennedy DO. Acute, dose-dependent cognitive effects of Ginkgo biloba, Panax ginseng and their combination in healthy young volunteers: differential interactions with cognitive demand. Hum Psychopharmacol. 2002 Jan;17(1):35-44. doi: 10.1002/hup.352. PMID 12404705
- [Background] Fekete M, Lehoczki A, Tarantini S, Fazekas-Pongor V, Csipo T, Csizmadia Z, Varga JT. Improving Cognitive Function with Nutritional Supplements in Aging: A Comprehensive Narrative Review of Clinical Studies Investigating the Effects of Vitamins, Minerals, Antioxidants, and Other Dietary Supplements. Nutrients. 2023 Dec 15;15(24):5116. doi: 10.3390/nu15245116. PMID 38140375
- [Background] Ping FW, Keong CC, Bandyopadhyay A. Effects of acute supplementation of Panax ginseng on endurance running in a hot & humid environment. Indian J Med Res. 2011 Jan;133(1):96-102. PMID 21321426
- [Background] Morris AC, Jacobs I, McLellan TM, Klugerman A, Wang LC, Zamecnik J. No ergogenic effect of ginseng ingestion. Int J Sport Nutr. 1996 Sep;6(3):263-71. doi: 10.1123/ijsn.6.3.263. PMID 8876346
- [Background] Engels HJ, Wirth JC. No ergogenic effects of ginseng (Panax ginseng C.A. Meyer) during graded maximal aerobic exercise. J Am Diet Assoc. 1997 Oct;97(10):1110-5. doi: 10.1016/S0002-8223(97)00271-X. PMID 9336557
- [Background] Allen JD, McLung J, Nelson AG, Welsch M. Ginseng supplementation does not enhance healthy young adults' peak aerobic exercise performance. J Am Coll Nutr. 1998 Oct;17(5):462-6. doi: 10.1080/07315724.1998.10718795. PMID 9791844
- [Background] Hsu CC, Ho MC, Lin LC, Su B, Hsu MC. American ginseng supplementation attenuates creatine kinase level induced by submaximal exercise in human beings. World J Gastroenterol. 2005 Sep 14;11(34):5327-31. doi: 10.3748/wjg.v11.i34.5327. PMID 16149140
- [Background] Kulaputana O, Thanakomsirichot S, Anomasiri W. Ginseng supplementation does not change lactate threshold and physical performances in physically active Thai men. J Med Assoc Thai. 2007 Jun;90(6):1172-9. PMID 17624213
- [Background] Reay JL, Kennedy DO, Scholey AB. The glycaemic effects of single doses of Panax ginseng in young healthy volunteers. Br J Nutr. 2006 Oct;96(4):639-42. PMID 17010221